CLINICAL TRIAL: NCT01625559
Title: A Phase I, Open-Label, Prospective Study to Determine the Safety and Tolerability of Sub-retinal Transplantation of Human Embryonic Stem Cell Derived Retinal Pigmented Epithelial(MA09-hRPE) Cells in Patients With Stargardt's Macular Dystrophy(SMD)
Brief Title: Safety and Tolerability of MA09-hRPE Cells in Patients With Stargardt's Macular Dystrophy(SMD)
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: CHABiotech CO., Ltd (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CHA_CTP_0903
Record Dates: First submitted 2012-06-18; First posted 2012-06-21 (Estimated); Last update posted 2024-04-10 (Actual); Status verified 2024-02

CONDITIONS: Stargardt's Macular Dystrophy

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- MA09-hRPE administration (Experimental): Biological: MA09-hRPE Cellular therapy
  Interventions: Biological: MA09-hRPE

INTERVENTIONS:
Biological: MA09-hRPE — MA09-hRPE cells

SUMMARY:
The purpose of this study is to evaluate the safety and tolerability of RPE cellular therapy in patients with SMD

DETAILED DESCRIPTION:
* to evaluate the safety and tolerability of RPE cellular therapy in patients with SMD
* to evaluate the preliminary efficacy of MA09-hPRE in patients with SMD

ELIGIBILITY:
Inclusion Criteria:

* Adult male or female over 20 years of age.
* Clinical diagnosis of advanced SMD.
* The visual acuity of the eye to receive the transplant will be no better than hand movement.
* The visual acuity of the eye that is not to receive the transplant will be no better than 24 (20/320) Early Treatment of Diabetic Retinopathy Study (ETDRS) letters.

Exclusion Criteria:

* History of malignancy.
* History of myocardial infarction in previous 12 months.
* History of diabetes mellitus.
* Any immunodeficiency.
* Any current immunosuppressive therapy other than intermittent or low dose cortico steroids.
* Serologic evidence of infection with Hepatitis B, Hepatitis C, or HIV.
* Current participation in any other clinical trial.
* Participation within previous 6 months in any clinical trial of a drug by ocular or systemic administration.
* Any other sight-threatening ocular disease.
* Any chronic ocular medications. Any history of retinal vascular disease (compromised blood-retinal barrier). Glaucoma. Uveitis or other intraocular inflammatory disease. Significant lens opacities or other media opacity. Ocular lens removal within previous 3 months

Min Age: 20 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 3 (Actual)
Dates: Start 2012-09; Primary Completion 2015-04 (Actual); Study Completion 2015-04 (Actual)

PRIMARY OUTCOMES:
safety and tolerance of transplantation | 18 months
  The transplantation of hESC-derived RPE cells MA09-hRPE will be considered safe and tolerated in the absence of:
  1. Any grade 2 (NCI grading system) or greater adverse event related to the cell product
  2. Any evidence that the cells are contaminated with an infectious agent
  3. Any evidence that the cells show tumorigenic potential

SECONDARY OUTCOMES:
Evidence of successful engraftment | 18 months
  Evidence of successful engraftmentEvidence of successful engraftment will consist of:
  Structural evidence (OCT imaging, fluorescein angiography, autofluorescense photography, slit-lamp examination with fundus photography) that cells have been implanted in the correct location Electroretinographic evidence (mfERG) showing enhanced activity in the implant location

CONTACTS AND LOCATIONS:
Overall Officials: Wonkyung Song, Principal Investigator — CHA Bundang Medical Center
Locations (1):
- CHA Bundang Medical Center, Seongnam-si, Gyeonggi-do, South Korea

REFERENCES:
- [Derived] Sung Y, Lee MJ, Choi J, Jung SY, Chong SY, Sung JH, Shim SH, Song WK. Long-term safety and tolerability of subretinal transplantation of embryonic stem cell-derived retinal pigment epithelium in Asian Stargardt disease patients. Br J Ophthalmol. 2021 Jun;105(6):829-837. doi: 10.1136/bjophthalmol-2020-316225. Epub 2020 Jul 29. PMID 32727729